CLINICAL TRIAL: NCT03698630
Title: Single Dose Oral Dexamethasone Versus Multi-dose Prednisolone in the Treatment of Acute Exacerbations of Asthma in Children Who Attend the Emergency Department
Brief Title: Single Dose Oral Dexamethasone Versus Multi-dose Prednisolone in the Treatment of Acute Exacerbations of Asthma in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: National Children's Research Centre (Unknown); Our Lady's Children's Hospital, Crumlin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESP_301_2010; 2010-022001-18 (EudraCT Number); ISRCTN26944158 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2018-09-11; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Asthma; Acute Asthma
Keywords: Asthma; Pediatric; Corticosteroid; Emergency department
MeSH Terms: conditions — Asthma; Emergencies | interventions — prednisolone phosphate; Methylprednisolone; Prednisolone; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, non-inferiority trial
Who Masked: Outcomes Assessor
Masking Description: The Pediatric Respiratory Assessment Measure score will be performed by a clinician blinded to treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Single dose of 0.3 mg/kg dexamethasone (rounded off to the nearest 2 mg, max. 12 mg) prescribed on day 1
  Interventions: Drug: Dexamethasone
- Prednisolone (Active Comparator): 1 mg/kg prednisolone (rounded off to the nearest 5 mg, max. 40 mg) prescribed daily for three days from day 1
  Interventions: Drug: Prednisolone Sodium Phosphate

INTERVENTIONS:
Drug: Prednisolone Sodium Phosphate — Prednesol 5mg Tablets (Phoenix Labs Ltd). Pink, circular, flat, bevel-edged scored tablets containing 5 mg of prednisolone as prednisolone sodium phosphate.
  Other Names: Prednesol 5mg; Prednisolone
  Arms: Prednisolone
Drug: Dexamethasone — Dexamethasone 2 mg tablets (Organon Ireland Ltd). Round, 6 mm, flat, white tablet with the code "XC/8" engraved on one surface and "Organon*" on the other containing 2 mg dexamethasone.
  Arms: Dexamethasone

SUMMARY:
A trial to investigate if a single dose of the oral corticosteroid, Dexamethasone is as effective in treating exacerbations of asthma in children as 3 days of treatment with another oral corticosteroid, Prednisolone

DETAILED DESCRIPTION:
Asthma is a major cause of pediatric morbidity and mortality. In acute exacerbations of asthma, corticosteroids reduce relapses, subsequent hospital admission and the need for ß2-agonist therapy. Prednisolone is relatively short-acting with a half-life of 12 to 36 hours, thereby requiring daily dosing. Prolonged treatment course, vomiting and a bitter taste may reduce patient compliance with prednisolone. Dexamethasone is a long-acting corticosteroid with a half-life of 36 to 72 hours. It is used frequently in children with croup and bacterial meningitis, and is well absorbed orally. The purpose of this trial is to examine whether a single dose of oral dexamethasone (0.3 mg/kg) is clinically non-inferior to prednisolone (1 mg/kg/day for three days) in the treatment of exacerbations of asthma in children who attend the Emergency Department.

This is a randomized, non-inferiority, open-label clinical trial. After informed consent with or without assent, patients will be randomized to either oral dexamethasone 0.3 mg/kg stat or prednisolone 1 mg/kg/day for three days. The primary outcome measure is the comparison between the Pediatric Respiratory Assessment Measure (PRAM) across both groups on Day 4. The PRAM score, a validated, responsive and reliable tool to determine asthma severity in children aged 2 to 16 years, will be performed by a clinician blinded to treatment allocation. Secondary outcomes include relapse, hospital admission and requirement for further steroid therapy. Data will be analyzed on an intention-to-treat and a per protocol basis. With a sample size of 232 subjects (105 in each group with an estimated 10% loss to follow-up), we will be able to reject the null hypothesis - that the population means of the experimental and control groups are equal with a power of 0.9. The Type I error probability associated with this test (of the null hypothesis) is 0.05.

This clinical trial may provide evidence that a shorter steroid course using dexamethasone can be used in the treatment of acute pediatric asthma, thus eliminating the issue of compliance to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 to 16 years
* Background history of asthma as defined by at least one previous episode of ß2-agonist-responsive wheeze in a child two years of age or over or a prior diagnosis of asthma, made by a pediatrician, or clinician of comparable experience
* Presentation with an asthma exacerbation as defined as acute asthma, which prompts assessment at the ED, and has any, or all, of the following clinical features: Dyspnea, Wheeze, Acute cough, Increased work of breathing, Increased requirement for ß2-agonist from baseline use or O2 saturation <95%

Exclusion Criteria:

* Less than 2 years old or over 16 years
* Critical or life-threatening asthma (as defined below)
* Known TB exposure
* Active varicella or herpes simplex infection
* Documented concurrent infection with RSV
* Fever >39.5°C
* Use of oral corticosteroids in the previous four weeks
* Concurrent stridor
* Galactose intolerance, the Lapp-lactase deficiency or glucose-galactose malabsorption
* Significant co-morbid disease: lung, cardiac, immune, liver, endocrine, neurological or psychiatric

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2012-07-13 (Actual); Study Completion 2012-07-13 (Actual)

PRIMARY OUTCOMES:
Pediatric Respiratory Assessment Measure score (PRAM) score | Day 4
  Pediatric Respiratory Assessment Measure score (PRAM) on Day 4. This is a compound score ranging from 0 to 12 that measures asthma severity by accounting for oxygen saturation, the presence of suprasternal retractions and/or Scalene muscle contractions, the degree of air entry and presence/type of wheezing.
  A score of 0-3 indicates mild asthma, 4-7 moderate asthma and 8-12 severe asthma.

SECONDARY OUTCOMES:
Relapse rate | 14 days
  Rate of relapse as defined as any visit to a healthcare provide as a result of asthma symptoms within 14 days of study enrollment
Salbutamol therapies | 14 days
  Frequency of salbutamol therapies given following enrolment
Compliance with medication as assessed by interview | 14 days
  Incidence of compliance with medication with regards to taking 3 doses of the medication.
Incidence of vomiting | 14 days
  Incidence of vomiting
Relapse rate | 14 days
  Relapse will be defined as any visit to a healthcare provider, for example, General Practitioner, ED, as a result of asthma symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Our Lady's Children's Hospital, Crumlin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cronin J, Kennedy U, McCoy S, An Fhaili SN, Crispino-O'Connell G, Hayden J, Wakai A, Walsh S, O'Sullivan R. Single dose oral dexamethasone versus multi-dose prednisolone in the treatment of acute exacerbations of asthma in children who attend the emergency department: study protocol for a randomized controlled trial. Trials. 2012 Aug 21;13:141. doi: 10.1186/1745-6215-13-141. PMID 22909281